CLINICAL TRIAL: NCT05149482
Title: Evolutionary Profile of Isolated Lateral Semicircular Canal Deficits on the Video Head Impulsed Test (VHIT)
Brief Title: Isolated Deficits of the Lateral Semicircular Canal
Acronym: CSL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8397
Record Dates: First submitted 2021-11-24; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Peripheral Vestibular Disorder
Keywords: Peripheral Vestibular Disorder; Lateral semicircular canal; Video Head Impulsed Test

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There are only a few cases of isolated lateral canal deficit described in the literature. This study would focus on this group of patients in order to establish an evolving profile, a recovery behavior that we could compare to that in the literature.

In addition, the evolving profile as well as the other clinical criteria identified would allow investigators to make hypotheses as to the pathology responsible for a given evolutionary profile.

The population studied is represented by adult patients admitted by the emergency consultation service of otolaryngology of the University Hospitals of Strasbourg for an acute unilateral vestibular deficit whose examination at the VHOT shows a reduced and isolated gain of a lateral semicircular canal.

ELIGIBILITY:
Inclusion criteria

* Major patient
* Man or woman
* Patient who has given their consent to the use of their data.
* Patient treated in the ENT department for dizziness between June 2020 and July 2021.

Non-inclusion criteria

* Patient who expressed his opposition to participating in the study
* Inability to provide the subject with enlightened information (difficulties in understanding the subject, cognitive disorders)
* Subject under safeguard of justice
* Subject under guardianship or guardianship
* Neurological signs on clinical examination

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient treated in the ENT department for dizziness between June 2020 and July 2021.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Establish the evolutionary profiles of patients with isolated lateral canal involvement | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Anne CHARPIOT, MD, PhD, Principal Investigator — Oto-rhino-laryngologie et Chirurgie cervico-faciale - Hôpitaux Universitaires de Strasbourg
Locations (1):
- Oto-rhino-laryngologie et Chirurgie cervico-faciale - Hôpitaux Universitaires de Strasbourg, Strasbourg, France